CLINICAL TRIAL: NCT00489216
Title: Weekly Subcutaneous Efalizumab for the Treatment of Steroid Refractory Graft-Versus-Host Disease of the Skin and Liver
Brief Title: Efalizumab in Treating Patients With Graft-Versus-Host Disease of the Skin That Did Not Respond to Previous Steroids
Acronym: NRR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient accrual/funding withdrawn
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC 0605
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Graft Versus Host Disease
Keywords: Graft Versus Host Disease; GVHD; Efalizumab; Raptiva; Steroid; Refractory; Skin; Liver; Lineberger; University of North Carolina
MeSH Terms: conditions — Graft vs Host Disease | interventions — efalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Efalizumab (Experimental): All patients on study will receive a total of 8 injections of efalizumab
  Interventions: Biological: efalizumab

INTERVENTIONS:
Biological: efalizumab — Efalizumab will be administered as a subcutaneous injection once a week for 8 weeks (total of 8 doses). First efalizumab injection will be dosed at 0.7mg/kg. Subsequent weekly injections given on days 8-50 will be dosed at
  1mg/kg
  Other Names: Raptiva

SUMMARY:
RATIONALE: Efalizumab may be an effective treatment for graft-versus-host disease of the skin caused by a donor stem cell transplant.

PURPOSE: This clinical trial is studying the side effects and how well efalizumab works in treating patients with graft-versus-host disease of the skin that did not respond to previous steroids.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the general safety of efalizumab in patients with cutaneous graft-vs-host disease (GVHD).
* Study the feasibility of digital imaging to objectively quantify cutaneous GVHD.
* Evaluate the feasibility of serial skin biopsies to monitor disease response to efalizumab in patients with cutaneous GVHD.

Secondary

* Assess the overall complete response rate in patients treated with this drug.
* Assess the overall cutaneous response rate (complete cutaneous response rate and partial cutaneous response rate) in patients treated with this drug.
* Assess the overall hepatic response rate (complete hepatic response rate and partial hepatic response rate) in patients treated with this drug.
* Assess the duration of any responses observed.
* Assess the effect of this drug on overall patient survival.
* Use the preliminary efficacy and toxicity data collected in this small exploratory study to decide on the appropriateness of a larger, subsequent phase II trial to more formally assess toxicity and efficacy of this drug in this patient population.
* Collect pharmacokinetic data on this drug in these patients.

OUTLINE: Patients receive efalizumab subcutaneously once weekly for 8 weeks (total of 8 doses).

Digital photographs of body regions are taken for determination of disease involved body surface area. Skin biopsies are obtained before and after treatment and analyzed for lymphocyte function associated antigen (LFA-1), intercellular adhesion molecule (ICAM-1), cluster of differentiation 4, 8, and possibly 20 (CD4, CD8, CD20) by immunohistochemistry.

After completion of study therapy, patients are followed at 1 and 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Skin disease

   * Patients must demonstrate evidence of an erythematous maculopapular rash which is felt to be clinically consistent with graft-versus-host disease. Patients must undergo skin biopsy prior to enrollment. Because the pathological findings of GVHD may be equivocal (6) a biopsy which is felt to be consistent with GVHD will be considered adequate.
   * Consider sclerodermatous skin changes may be present but will not by themselves adequate for enrollment. Patients must exhibit signs of an active inflammatory rash.
2. Liver disease

   • Although hepatic involvement is not required for study participation, patients with concomitant GVHD of the liver are encouraged to enroll. All patients with hepatic GVHD must also demonstrate cutaneous disease. Patients with liver dysfunction are encouraged but not required to undergo hepatic biopsy in order to document that liver injury is the result of GVHD. Patients with a pretreatment serum bilirubin ≥ 2.0 mg/dL and biopsy-confirmed cutaneous GVHD will be assumed to demonstrate hepatic GVHD if no other cause for the liver function test (LFT) elevation can be identified.
3. Age ≥ 18 years
4. Patients must be ≥ 30 days removed from allogeneic hematopoietic stem cell transplant in order to allow for engraftment. Patients receiving peripheral blood stem cells and/or bone marrow will be eligible, regardless of the degree of human leukocyte antigen (HLA) matching.
5. Steroid refractory disease

   • All patients must demonstrate evidence of steroid refractory graft-versus host disease of the skin or liver. In an effort to conform to a standard definition of steroid refractory disease, we will base our criteria on those described in a large intergroup trial examining the effectiveness of pentostatin for steroid refractory chronic GVHD (31). Because the present study, however, is designed to include patients with both acute and chronic GVHD based on traditional disease classification criteria, the required time intervals necessary to define steroid-refractoriness have been shortened. Patients will be considered steroid refractory if any one of the following conditions is met:
   * Worsening skin or liver disease despite 1 week on the equivalent of 1mg/kg of methylprednisolone
   * Failure to achieve a 50% reduction in the body surface area involved by GVHD or a 50% reduction in the total serum bilirubin after 4 weeks on the equivalent of at least 0.5 mg/kg of methylprednisolone
   * Requirement of ≥ the equivalent of 0.5mg/kg of methylprednisolone to maintain a response after 8 weeks of steroid therapy
   * Patients with progression of cutaneous or hepatic GVHD after a prior history of treatment with at least 8 weeks of corticosteroids now requiring the reintroduction of corticosteroids (> the equivalent of 10mg/day of methylprednisolone)
   * Patients with GVHD not improving or progressing on alternative immunosuppressive agents will be eligible if steroid refractoriness has been established previously
6. Required initial laboratory values:

Absolute neutrophil count (ANC) > 1000/μL Platelet count ≥ 20,000/μL Serum creatinine ≤ 3.0 mg/dL

Exclusion Criteria:

1. Non-pregnant and non-nursing

   • Treatment under this protocol would expose an unborn child to significant risks. Women and men of reproductive potential must agree to use an effective means of birth control.
2. No HIV infection

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 2 terminal half-lives since prior and no concurrent infliximab, daclizumab, etanercept, rituximab, antithymocyte globulin (ATG), or denileukin diftitox

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-12; Primary Completion 2008-06 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C. Shea, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://clinicaltrials.gov/ct2/show/NCT00489216?term=LCCC0605&rank=1

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients with evidence of an inflammatory, erythematous rash and skin biopsy consistent with cutaneous Graft-Versus-Host disease who had failed to improve after at least 4 weeks of methylprednisolone at 0.5mg/kg were eligible for enrollment.
Groups:
- Efalizumab: All patients on study will receive a total of 8 injections of efalizumab
  efalizumab: Efalizumab will be administered as a subcutaneous injection once a week for 8 weeks (total of 8 doses). First efalizumab injection will be dosed at 0.7mg/kg. Subsequent weekly injections given on days 8-50 will be dosed at
  1mg/kg
Period: Overall Study
Arm/Group | Efalizumab
Started | 2
Completed | 1
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Patients with evidence of an inflammatory, erythematous rash and skin biopsy consistent with cutaneous Graft-Versus-Host disease who had failed to improve after at least 4 weeks of methylprednisolone at 0.5mg/kg were eligible for enrollment. Two patients were enrolled in the study.
Arm/Group | Efalizumab
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Experiencing Adverse Events
Description: The primary objective of this exploratory study is to evaluate the general tolerability of efalizumab in patients suffering from steroid refractory GVHD
  Subjects will be evaluated for drug toxicity each visit. Toxicity will be graded using the Common Terminology Criteria for Adverse Events (CTCAE) common criteria.
Time Frame: 120 days
Population: Of the two patients, one patient completed all 8 doses of study medication according to schedule. The other patient received 6/8 scheduled efalizumab doses, but was subsequently taken off the study after developing transient coagulase negative staphylococcal bacteremia.
Measure: Number; unit: participants
Arm/Group | Efalizumab
Number analyzed (Participants) | 2
participants | 2

2. Primary Outcome: Degree of Skin Involvement by GVHD Using Two Digital Photography Techniques.
Description: Estimate of the percentage of body surface area involved by GVHD using two digital photography techniques and computerized image analyses:
  1. Digital photography and body surface area calculations: A total of 12 digital photographs were obtained from different body regions using systematic digital imaging and computerized image analysis.
  2. Body surface area calculations: Using National Institutes of Health image software, each body region will be manually traced and the total area of the traced area determined. Using a similar technique, each part of the region that is involved by a GVHD rash will also be traced and its area measured. The areas involved by rash will then be summed, and finally divided by the total area of the region. In so doing, the percentage of each region that is involved by GVHD will be determined.
Time Frame: 120 days
Population: Data was not collected for this objective due to limited number of participants. A minimum of 12 patients were needed for analysis.
Arm/Group | Efalizumab
Number analyzed (Participants) | 0

3. Primary Outcome: Exploratory Assessment of the Staining of Cutaneous Tissues for LFA-1, ICAM-1, CD4, CD8, and Possibly CD20
Description: Numerical scoring system for both LFA-1 and ICAM-1 expression which could then be used in a larger phase II trial to correlate clinical response rates to pathological findings.
Time Frame: 57 days
Population: There is no data for this outcome measure because of the small number of patients and inability to make meaningful conclusions
Arm/Group | Efalizumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Complete Response Rate
Description: To assess the overall complete response rate on study days 29 and 57 after 4 and 8 doses of weekly subcutaneous efalizumab. A complete response (CR) was defined as the total resolution of skin disease, and a partial response was defined as >=50% reduction in the proportion of total body surface area involved by rash.
Time Frame: 57 days
Population: Of the two patients, one patient completed all 8 doses of study medication according to schedule. The other patient received 6/8 scheduled efalizumab doses, but was subsequently taken off the study after developing transient coagulase negative staphylococcal bacteremia. The patient demonstrated a complete response (CR).
Measure: Count of Participants; unit: Participants
Arm/Group | Efalizumab
Number analyzed (Participants) | 2
Participants | 1

5. Secondary Outcome: Complete Cutaneous Response Rate
Description: The complete disappearance of all signs of cutaneous graft-versus-host disease. Complete cutaneous response rate + partial cutaneous response rate
Time Frame: On study days 29 and 57 after 4 and 8 doses of weekly subcutaneous efalizumab
Measure: Number; unit: participants
Arm/Group | Efalizumab
Number analyzed (Participants) | 2
participants | 1

6. Secondary Outcome: Overall Hepatic Response Rate
Description: The normalization of the total serum bilirubin to <2mg/dL
Time Frame: On study days 29 and 57 after 4 and 8 doses of weekly subcutaneous efalizumab
Population: There is no data for this outcome measure as no enrolled patients had an elevated bilirubin level.
Arm/Group | Efalizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Final efalizumab dose administered on day 57. Patients observed for 8 additional weeks.
Arm/Group | Efalizumab
All-Cause Mortality (participants affected / at risk) | 1/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Efalizumab (N=2)
Transient Coagulase Negative Staphylococcal Bacteremia (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Efalizumab (N=2)
Nausea (Gastrointestinal disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to funding withdrawal/insufficient accrual limiting the data to be analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes